CLINICAL TRIAL: NCT04510194
Title: COVID-OUT: Early Outpatient Treatment for SARS-CoV-2 Infection (COVID-19)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: UnitedHealth Group (Industry); Northwestern University (Other); Hennepin County Medical Center, Minneapolis (Other); University of Colorado, Denver (Other); Olive View-UCLA Education & Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GIM-2020-29324
Record Dates: First submitted 2020-08-07; First posted 2020-08-12 (Actual); Results first posted 2023-07-13 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Covid19; SARS-CoV Infection
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Metformin; Fluvoxamine; Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the investigational pharmacy and unblinded statistician have access to patient treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment Arm - Metformin Only Group (Experimental): Participants in the treatment arm of the trial are those who test positive for SARS-COV-2 infection at the time of screening. Participants in this arm and group will receive the metformin alone.
  Interventions: Drug: Metformin
- Treatment Arm - Placebo Group (Placebo Comparator): Participants in the treatment arm of the trial are those who test positive for SARS-COV-2 infection at the time of screening. Participants in this arm and group will receive the placebo.
  Interventions: Drug: Placebo
- Treatment Arm - Ivermectin Only Group (Experimental): Participants in the treatment arm of the trial are those who test positive for SARS-COV-2 infection at the time of screening. Participants in this arm and group will receive the ivermectin alone.
  Interventions: Drug: Ivermectin
- Treatment Arm - Fluvoxamine Only Group (Experimental): Participants in the treatment arm of the trial are those who test positive for SARS-COV-2 infection at the time of screening. Participants in this arm and group will receive the fluvoxamine alone.
  Interventions: Drug: Fluvoxamine
- Treatment Arm - Metformin and Fluvoxamine Group (Experimental): Participants in the treatment arm of the trial are those who test positive for SARS-COV-2 infection at the time of screening. Participants in this arm and group will receive metformin and fluvoxamine.
  Interventions: Drug: Metformin; Drug: Fluvoxamine
- Treatment Arm - Metformin and Ivermectin Group (Experimental): Participants in the treatment arm of the trial are those who test positive for SARS-COV-2 infection at the time of screening. Participants in this arm and group will receive metformin and ivermectin.
  Interventions: Drug: Metformin; Drug: Ivermectin

INTERVENTIONS:
Drug: Metformin — Metformin; immediate release formation; 500mg on Day 1; 500mg BID on Day 2 through Day 5; 500mg in AM and 1,000mg in PM on Day 6 through Day 14.
  Other Names: glucophage
  Arms: Treatment Arm - Metformin Only Group; Treatment Arm - Metformin and Fluvoxamine Group; Treatment Arm - Metformin and Ivermectin Group
Drug: Placebo — placebo; appearance and size are exact matching to the three study drugs.
  Arms: Treatment Arm - Placebo Group
Drug: Fluvoxamine — An antidepressant, administered 50mg per day on Day 1; then 50mg twice-daily for Day 2 through Day 14
  Other Names: Luvox
  Arms: Treatment Arm - Fluvoxamine Only Group; Treatment Arm - Metformin and Fluvoxamine Group
Drug: Ivermectin — An anti-parasitic medication administered as 390mcg/kg to 470mcg/kg per day for 3 days
  Other Names: Stromectol
  Arms: Treatment Arm - Ivermectin Only Group; Treatment Arm - Metformin and Ivermectin Group

SUMMARY:
The purpose of this trial is to understand whether:

1. Metformin vs fluvoxamine vs ivermectin vs metformin+fluvoxamine vs metformin+ivermectin is superior to placebo in non-hospitalized adults with SARS-CoV-2 disease for preventing Covid-19 disease progression.
2. To understand if the active treatment arms are superior to placebo in improving viral load, serologic markers associated with Covid-19, and gut microbiome in non-hospitalized adults with SARS-CoV-2 infection.
3. To understand if any of the active treatment arms prevent long-covid syndrome, PASC (post-acute sequelae of SARS-CoV-2 infection).

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is a rapidly spreading viral infection causing COVID-19 disease. There currently is no definitive preventive or early outpatient treatment therapy for Covid-19. Study study assess 3 existing generic medications: metformin, fluvoxamine, and ivermectin.

Metformin: in-silico, in-vitro, ex-vivo tissue assays suggest that metformin inhibits viral replication of SARS-CoV-2 virus (Castle et al; Gordon et al; and Schaller et al). Several retrospective cohort analyses have suggested an association between taking metformin prior to SARS-CoV-2 infection and less severe outcomes. Kow, J Med Virol conducted a meta analysis, with an overall odds ratio for mortality of 0.62 (0.43-0.89). Gordon et al found decreased SARS-CoV-2 and increased cell viability with metformin in vitro. (Gordon et al, Nature). While anti-viral activity may be contributing to the observational associations of reduced severity of Covid-19, metformin has a proven history of beneficial immune-modulatory effects, including on CRP, IL-6 and TNF-alpha, neutrophil extracellular traps, and improved T cell immunity. Outpatient metformin use has now been associated with lower IL-6, CRP, and neutrophil-lymphocyte ratio in persons with Covid-19 (Lou et al, Diabetes Care 2020).

Fluvoxamine: appears to have anti-inflammatory effects in SARS-CoV-2 infection. There is evidence that SARS-CoV-2 infection causes ER stress and activates pathways of unfolded protein response. Sigma-1 receptor (S1R) is an ER chaperone protein that regulates cytokine production through interaction with IRE1. Fluvoxamine is a selective serotonin reuptake inhibitor that is a powerful S1R agonist. Fluvoxamine has previously been shown to protect mice from septic shock and reduce the inflammatory response. There is potential for fluvoxamine as an immunomodulatory treatment for SARS-Cov-2. Fluvoxamine in CACO2 cells infected with SARS-Cov-2 had a reduction in production of a subset of cytokines including IL-6, IL-8, CXCL1, and CXCL10.53 A randomized controlled clinical trial of 152 patients showed that patients who received fluvoxamine were less likely to experience clinical deterioration, or serious adverse events due to SARS-Cov-2 when compared to placebo (0% vs. 8%). A follow-up real-world observational cohort had similar findings of 0% (0/65) hospitalization with fluvoxamine vs. 12% (6/48) with observation.

Ivermectin has also shown anti-inflammatory effects that would reduce the harmful cytokine cascade noted in severe Covid-19 disease. A recent trial assessing a multi-therapy including 12mg one-time dose of ivermectin found a 75% reduction in hospitalizations. Another small double-blinded RCT showed significant increased chance of viral clearance after a 5-day course of ivermectin. Another March 2021 RCT reported no effect on diminishing symptoms, but was under-powered for assessing reductions in hospitalization. An RCT with ivermectin must be done in the US, as endemic strongyloidiasis in other countries may confound results.

Statistical Considerations:

An independent data safety monitoring board will assess safety approximately twice per month; and will assess futility and efficacy at least twice throughout the study. If one of the arms reaches pre-specified boundaries for futility or efficacy, the DSMB will recommend closing of that arm(s). The detailed statistical analysis plan will be developed by the blinded statistician and co-investigators and per the protocol will be submitted to the DSMB.

ELIGIBILITY:
Inclusion Criteria:

* Positive laboratory test for active SARS-CoV-2 viral infection based on local laboratory standard (i.e. +PCR) within 3 days of randomization.
* No known history of confirmed SARS-CoV-2 infection
* BMI >= 25kg/m2 by self-report height/weight or >= 23kg/m2 in patients who self-identify in South Asian or Latinx background.
* Willing and able to comply with study procedures (i.e. swallow pills)
* Has an address and electronic device for communication
* GFR>45ml/min within 2 weeks for patients >75 years old, or with history of heart, kidney, or liver failure.

Exclusion Criteria:

* Hospitalized, for COVID-19 or other reasons.
* Symptom onset greater than 7 days before randomization (symptoms not required for inclusion).
* Immune compromised state (solid organ transplant, bone marrow transplant, AIDS, on high dose steroids)
* Hepatic impairment (Child-Pugh B and C) or other condition that, in the opinion of the investigator, would affect safety
* Inability to obtain informed consent
* Enrollment in another blinded Randomized Controlled Trial for COVID-19
* Already received an effective (FDA approved/EUA*) therapy for COVID-19 (currently monoclonal antibody treatment)
* Alcohol use disorder
* Other unstable medical condition or combination of home medications that in the view of the PI make it unsafe for the individual to participate
* History of severe kidney disease i.e.:

  1. Stage 4 or 5 CKD, or Estimated Glomerular Filtration Rate (eGFR) of < 45ml/min/1.73 m2
  2. Other kidney disease that in the opinion of the investigator would affect clearance
* Unstable heart failure (Stage 3 or 4 heart failure)
* Allergic reaction to metformin, fluvoxamine, or ivermectin in the past
* Bipolar disease: individuals who report they have bipolar disorder or are taking medication for bipolar disorder (lithium, valproate, high-dose antipsychotic), unless the investigator concludes that the risk for mania is unlikely
* Current loa loa or onchocerciasis infection
* Typhoid, BCG, or cholera vaccination within the 14-days or 3 days after

Medication Exclusions:

* Cimetidine, hydroxychloroquine, insulin, sulfonylurea, dolutegravir, patiromer, ranolazine, tafenoquine.
* Rasagiline, selegiline, or monoamine oxidase inhibitors, linezolid, methadone
* Duloxetine, methylene blue
* Tizanidine, ramelteon, sodium picosulfate
* Alosetron, agomelatine, bromopride, dapoxetine, tamsimelteon, thioridazine, urokinase, pimozide

The following medications may not need to be excluded when dose for that individual is considered alongside the low dose of fluvoxamine being used and other medications being used. The PI or site PI may review and decide if the patient should be excluded from the fluvoxamine arms:

1. Taking SSRIs, SNRIs, or tricyclic antidepressants, unless these are at a low dose such that a study investigator concludes that a clinically significant interaction with fluvoxamine (ie either serotonin syndrome or TCA overdose) is unlikely (examples: participant takes escitalopram but only at 10mg daily; that dose plus 100mg fluvoxamine would be insufficient to cause serotonin syndrome; or, participant takes amitriptyline but only at 25mg nightly; even if fluvoxamine inhibits its metabolism, it would be an insufficient dose to cause QTc prolongation or problematic side effects). Risk Class C, monitor therapy.
2. Individuals who take alprazolam or diazepam and are unwilling to cut the medication by 20% (rationale: fluvoxamine modestly inhibits the metabolism of these drugs). Risk Class C, monitor therapy
3. Participants taking theophylline, clozapine, or olanzapine (drugs with a narrow therapeutic index that are primarily metabolized by CYP 1A2, which is inhibited by fluvoxamine) will be reviewed with a study investigator and excluded unless the investigator concludes that the risk to the participant is low (this would be unlikely; example: participant takes clozapine only as needed and is willing to avoid it for the 14 days of the study).
4. Patients will be advised that there is a small risk that the following substances will be affected by fluvoxamine, but that significant effects are not likely at the low dose being used: caffeine, nicotine, melatonin. Risk Class C, monitor therapy
5. Taking warfarin-also known as Coumadin, NSAIDs, and Aspirin (rationale: increased risk of bleeding), phenytoin (rationale: fluvoxamine inhibits its metabolism), clopidogrel (rationale: fluvoxamine inhibits its metabolism from pro-drug to active drug which raises risk of cardiovascular events), and St John's wort (rationale: fluvoxamine + St John's wort are considered contraindicated because of the risk of serotonin syndrome) Risk C, monitor therapy.

   * Additional COVID-19 treatments to exclude will be decided by a panel of at least 3 Co-Investigators on this study. The additional treatments to exclude will be documented and submitted to the IRB but may be implemented before formal IRB approval is complete. We take this approach because of the rapidly changing treatment landscape of COVID-19. Participation in the study does not prevent them from receiving such treatments after enrollment.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1323 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Bramante, MD, Principal Investigator — University of Minnesota
Locations (7):
- United States (7):
  - Olive View UCLA Medical Center, Sylmar, California
  - University of Colorado Denver; Department of Medicine; Anschutz Health and Wellness Center, Aurora, Colorado
  - New West Physicians, Golden, Colorado
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - American Health Network of Indiana, Greenfield, Indiana
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gordon DE, Jang GM, Bouhaddou M, Xu J, Obernier K, White KM, O'Meara MJ, Rezelj VV, Guo JZ, Swaney DL, Tummino TA, Huttenhain R, Kaake RM, Richards AL, Tutuncuoglu B, Foussard H, Batra J, Haas K, Modak M, Kim M, Haas P, Polacco BJ, Braberg H, Fabius JM, Eckhardt M, Soucheray M, Bennett MJ, Cakir M, McGregor MJ, Li Q, Meyer B, Roesch F, Vallet T, Mac Kain A, Miorin L, Moreno E, Naing ZZC, Zhou Y, Peng S, Shi Y, Zhang Z, Shen W, Kirby IT, Melnyk JE, Chorba JS, Lou K, Dai SA, Barrio-Hernandez I, Memon D, Hernandez-Armenta C, Lyu J, Mathy CJP, Perica T, Pilla KB, Ganesan SJ, Saltzberg DJ, Rakesh R, Liu X, Rosenthal SB, Calviello L, Venkataramanan S, Liboy-Lugo J, Lin Y, Huang XP, Liu Y, Wankowicz SA, Bohn M, Safari M, Ugur FS, Koh C, Savar NS, Tran QD, Shengjuler D, Fletcher SJ, O'Neal MC, Cai Y, Chang JCJ, Broadhurst DJ, Klippsten S, Sharp PP, Wenzell NA, Kuzuoglu-Ozturk D, Wang HY, Trenker R, Young JM, Cavero DA, Hiatt J, Roth TL, Rathore U, Subramanian A, Noack J, Hubert M, Stroud RM, Frankel AD, Rosenberg OS, Verba KA, Agard DA, Ott M, Emerman M, Jura N, von Zastrow M, Verdin E, Ashworth A, Schwartz O, d'Enfert C, Mukherjee S, Jacobson M, Malik HS, Fujimori DG, Ideker T, Craik CS, Floor SN, Fraser JS, Gross JD, Sali A, Roth BL, Ruggero D, Taunton J, Kortemme T, Beltrao P, Vignuzzi M, Garcia-Sastre A, Shokat KM, Shoichet BK, Krogan NJ. A SARS-CoV-2 protein interaction map reveals targets for drug repurposing. Nature. 2020 Jul;583(7816):459-468. doi: 10.1038/s41586-020-2286-9. Epub 2020 Apr 30. PMID 32353859
- [Background] Castle, B.T., C. Dock, M. Hemmat, S. Kline, C. Tignanelli, R. Rajasingham, D. Masopust, P. Provenzano, R. Langlois, T. Schacker, A. Haase, and D.J. Odde, Biophysical modeling of the SARS-CoV-2 viral cycle reveals ideal antiviral targets. bioRxiv, 2020. https://www.biorxiv.org/content/10.1101/2020.05.22.111237v2.
- [Derived] Hartman KM, Patel B, Rao V, Hagen AA, Saveraid HG, Fricton R, Lee S, Snyder AT, Pullen MF, Boulware DR, Liebovitz DM, Belani HK, Niklas JM, Murray TA, Cohen K, Thompson JL, Erickson SM, Bramante CT. A Comparison of Recruitment Methods for a Remote, Nationwide Clinical Trial for COVID-19 Treatment. Open Forum Infect Dis. 2024 Apr 29;11(7):ofae224. doi: 10.1093/ofid/ofae224. eCollection 2024 Jul. PMID 38947738
- [Derived] Bramante CT, Beckman KB, Mehta T, Karger AB, Odde DJ, Tignanelli CJ, Buse JB, Johnson DM, Watson RHB, Daniel JJ, Liebovitz DM, Nicklas JM, Cohen K, Puskarich MA, Belani HK, Siegel LK, Klatt NR, Anderson B, Hartman KM, Rao V, Hagen AA, Patel B, Fenno SL, Avula N, Reddy NV, Erickson SM, Fricton RD, Lee S, Griffiths G, Pullen MF, Thompson JL, Sherwood NE, Murray TA, Rose MR, Boulware DR, Huling JD; COVID-OUT Study Team. Favorable Antiviral Effect of Metformin on SARS-CoV-2 Viral Load in a Randomized, Placebo-Controlled Clinical Trial of COVID-19. Clin Infect Dis. 2024 Aug 16;79(2):354-363. doi: 10.1093/cid/ciae159. PMID 38690892
- [Derived] Bramante CT, Buse JB, Liebovitz DM, Nicklas JM, Puskarich MA, Cohen K, Belani HK, Anderson BJ, Huling JD, Tignanelli CJ, Thompson JL, Pullen M, Wirtz EL, Siegel LK, Proper JL, Odde DJ, Klatt NR, Sherwood NE, Lindberg SM, Karger AB, Beckman KB, Erickson SM, Fenno SL, Hartman KM, Rose MR, Mehta T, Patel B, Griffiths G, Bhat NS, Murray TA, Boulware DR; COVID-OUT Study Team. Outpatient treatment of COVID-19 and incidence of post-COVID-19 condition over 10 months (COVID-OUT): a multicentre, randomised, quadruple-blind, parallel-group, phase 3 trial. Lancet Infect Dis. 2023 Oct;23(10):1119-1129. doi: 10.1016/S1473-3099(23)00299-2. Epub 2023 Jun 8. PMID 37302406
- [Derived] Boulware DR, Murray TA, Proper JL, Tignanelli CJ, Buse JB, Liebovitz DM, Nicklas JM, Cohen K, Puskarich MA, Belani HK, Siegel LK, Klatt NR, Odde DJ, Karger AB, Ingraham NE, Hartman KM, Rao V, Hagen AA, Patel B, Fenno SL, Avula N, Reddy NV, Erickson SM, Lindberg S, Fricton R, Lee S, Zaman A, Saveraid HG, Tordsen WJ, Pullen MF, Sherwood NE, Huling JD, Bramante CT; COVID-OUT study team. Impact of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Vaccination and Booster on Coronavirus Disease 2019 (COVID-19) Symptom Severity Over Time in the COVID-OUT Trial. Clin Infect Dis. 2023 Feb 8;76(3):e1-e9. doi: 10.1093/cid/ciac772. PMID 36124697
- [Derived] Bramante CT, Huling JD, Tignanelli CJ, Buse JB, Liebovitz DM, Nicklas JM, Cohen K, Puskarich MA, Belani HK, Proper JL, Siegel LK, Klatt NR, Odde DJ, Luke DG, Anderson B, Karger AB, Ingraham NE, Hartman KM, Rao V, Hagen AA, Patel B, Fenno SL, Avula N, Reddy NV, Erickson SM, Lindberg S, Fricton R, Lee S, Zaman A, Saveraid HG, Tordsen WJ, Pullen MF, Biros M, Sherwood NE, Thompson JL, Boulware DR, Murray TA; COVID-OUT Trial Team. Randomized Trial of Metformin, Ivermectin, and Fluvoxamine for Covid-19. N Engl J Med. 2022 Aug 18;387(7):599-610. doi: 10.1056/NEJMoa2201662. PMID 36070710
- [Derived] Dodds MG, Doyle EB, Reiersen AM, Brown F, Rayner CR. Fluvoxamine for the treatment of COVID-19. Lancet Glob Health. 2022 Mar;10(3):e332. doi: 10.1016/S2214-109X(22)00006-7. No abstract available. PMID 35180412

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm - Metformin Only Group | Treatment Arm - Placebo Group | Treatment Arm - Ivermectin Only Group | Treatment Arm - Fluvoxamine Only Group | Treatment Arm - Metformin and Fluvoxamine Group | Treatment Arm - Metformin and Ivermectin Group
Started | 284 | 295 | 206 | 159 | 175 | 204
Completed | 278 | 291 | 206 | 156 | 173 | 201
Not Completed | 6 | 4 | 0 | 3 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm - Metformin Only Group | Treatment Arm - Placebo Group | Treatment Arm - Ivermectin Only Group | Treatment Arm - Fluvoxamine Only Group | Treatment Arm - Metformin and Fluvoxamine Group | Treatment Arm - Metformin and Ivermectin Group | Total
Number analyzed (Participants) | 284 | 295 | 206 | 159 | 175 | 204 | 1323
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 46 [36 to 56] | 42 [36 to 54] | 48 [39 to 57] | 46 [38 to 53] | 46 [38 to 53] | 46 [39 to 53] | 46 [37 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 187 | 108 | 87 | 83 | 108 | 741
  Male | 116 | 108 | 98 | 72 | 92 | 96 | 582
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 4 | 4 | 1 | 1 | 18
  Asian | 7 | 9 | 6 | 5 | 4 | 7 | 38
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 0 | 1 | 1 | 5
  Black or African American | 20 | 15 | 12 | 13 | 14 | 13 | 87
  White | 213 | 238 | 151 | 125 | 141 | 154 | 1022
  More than one race | 10 | 4 | 5 | 4 | 2 | 5 | 30
  Unknown or Not Reported | 29 | 23 | 28 | 8 | 12 | 23 | 123

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Hypoxia Only
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm - Metformin Only Group | Treatment Arm - Placebo Group | Treatment Arm - Ivermectin Only Group | Treatment Arm - Fluvoxamine Only Group | Treatment Arm - Metformin and Fluvoxamine Group | Treatment Arm - Metformin and Ivermectin Group
Number analyzed (Participants) | 278 | 291 | 206 | 156 | 173 | 201
Participants | 147 | 158 | 88 | 73 | 71 | 96

2. Primary Outcome: Count of Participants With ED Visit, Hospitalization or Death
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm - Metformin Only Group | Treatment Arm - Placebo Group | Treatment Arm - Ivermectin Only Group | Treatment Arm - Fluvoxamine Only Group | Treatment Arm - Metformin and Fluvoxamine Group | Treatment Arm - Metformin and Ivermectin Group
Number analyzed (Participants) | 278 | 291 | 206 | 156 | 173 | 201
Participants | 27 | 48 | 16 | 15 | 18 | 23

3. Primary Outcome: Count of Participants With Hospitalization or Death
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm - Metformin Only Group | Treatment Arm - Placebo Group | Treatment Arm - Ivermectin Only Group | Treatment Arm - Fluvoxamine Only Group | Treatment Arm - Metformin and Fluvoxamine Group | Treatment Arm - Metformin and Ivermectin Group
Number analyzed (Participants) | 278 | 291 | 206 | 156 | 173 | 201
Participants | 8 | 18 | 5 | 5 | 6 | 4

4. Primary Outcome: Count of Participants Who Died
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm - Metformin Only Group | Treatment Arm - Placebo Group | Treatment Arm - Ivermectin Only Group | Treatment Arm - Fluvoxamine Only Group | Treatment Arm - Metformin and Fluvoxamine Group | Treatment Arm - Metformin and Ivermectin Group
Number analyzed (Participants) | 278 | 291 | 206 | 156 | 173 | 201
Participants | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Treatment Arm - Metformin Only Group | Treatment Arm - Placebo Group | Treatment Arm - Ivermectin Only Group | Treatment Arm - Fluvoxamine Only Group | Treatment Arm - Metformin and Fluvoxamine Group | Treatment Arm - Metformin and Ivermectin Group
All-Cause Mortality (participants affected / at risk) | 0/284 | 0/295 | 0/206 | 0/159 | 0/175 | 1/204
Serious Adverse Events (participants affected / at risk) | 0/284 | 0/295 | 0/206 | 0/159 | 0/175 | 0/204
Other Adverse Events (participants affected / at risk) | 0/284 | 2/295 | 1/206 | 0/159 | 0/175 | 0/204
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm - Metformin Only Group (N=284) | Treatment Arm - Placebo Group (N=295) | Treatment Arm - Ivermectin Only Group (N=206) | Treatment Arm - Fluvoxamine Only Group (N=159) | Treatment Arm - Metformin and Fluvoxamine Group (N=175) | Treatment Arm - Metformin and Ivermectin Group (N=204)
neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dizziness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
weakness in leg/arms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT04510194/Prot_SAP_001.pdf